CLINICAL TRIAL: NCT07167212
Title: Comparative Effect of Diaphragmatic Training and Myofascial Release on Pain Flexibility and Disability in Patients With Chronic Non-specific Low Back Pain
Brief Title: Comparative Effect of Diaphragmatic Training in Patients With Chronic Non-specific Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This record is a duplicate of IRCT20220604055072N3, where the trial was prospectively registered. Entered here in error.
Sponsor: Rashid Latif Medical College (Other)
Responsible Party: Principal Investigator, Aleena Waheed, Senior Lecturer, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2024/213
Record Dates: First submitted 2025-09-01; First posted 2025-09-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non Specific Low Back Pain
Keywords: Pain; Flexibility; Disability; Strength; Lumbar
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm Training (Experimental): Diaphragm Training
  Interventions: Other: Diaphragm Training
- Myofascial Release technique (Active Comparator): Myofascial Release technique
  Interventions: Other: Myofascial Release Technique

INTERVENTIONS:
Other: Diaphragm Training — The diaphragm serves dual roles in respiration and postural control, yet its contribution is often overlooked in core stability exercise (CSE) programs for low back pain (LBP) rehabilitation. Abdominal hollowing, or the 'tummy tuck,' targets TrA and lumbar multifidus. Diaphragmatic breathing (DB) increases intra-abdominal pressure, contributing to lumbar stability. The intervention included four progressive weeks: Week 1-Supine and Crocodile breathing; Week 2-Supine and Crocodile with TheraBand; Week 3-Seated and 90/90/90 breathing; Week 4-Seated and 90/90/90 with TheraBand. Supine emphasized diaphragmatic expansion with resistance at the thoracolumbar junction; Crocodile focused on lateral rib expansion; Seated required upright posture with rib control; 90/90/90 integrated deep breathing with resisted stabilization. This study evaluates DB combined with CSE on pain, disability, muscle activity, and sleep quality in chronic LBP.
  Arms: Diaphragm Training
Other: Myofascial Release Technique — The myofascial release technique for the diaphragm was performed with the participant lying supine and limbs relaxed. The therapist, positioned at the head, placed the pisiform, hypothenar, and last three fingers bilaterally under the seventh to tenth rib costal cartilages, forearms aligned toward the shoulders. During inspiration, gentle traction was applied cephalad and slightly laterally, accompanying rib elevation. On exhalation, pressure was directed inward along the costal margin to maintain resistance. With each breath, traction was gradually deepened to improve release. The maneuver consisted of two sets of 10 deep breaths with a 1-minute rest between sets. Figure 1 illustrates the manual diaphragm release technique (source: author's photo). This method, adapted from Rocha et al. (2015), emphasizes progressive traction and controlled resistance to facilitate diaphragmatic mobility and rib cage expansion.
  Arms: Myofascial Release technique

SUMMARY:
Background: The diaphragm muscle is a respiratory muscle with postural function. Patients with chronic LBP (CLBP) are more susceptible to diaphragm fatigue than healthy people and, therefore, can likely benefit from exercises designed to improve strength/endurance in this muscle. Studying the results of diaphragmatic training versus myofascial release was a strategy for determining which of them was the most effective in improving pain, flexibility and disability in the patients with chronic non- specific low back pain.

Objective: The objective of the study will be to compare the effect of Diaphragm training and myofascial release back pain patients.

Methods: A randomized clinical trial will be conducted on 44 patients aged 20-45 years. The patients will be randomized using lottery method. Group A will underwent diaphragmatic training with four positions with hot-pack and therapeutic ultrasound as baseline treatment NPRS will be used to measure the intensity of pain, ODI for the measurement of disability and Schober's test for lumbar flexibility before and after the completion of treatment sessions. Group B will receive myofascial release of diaphragm for 15 minutes with two sets of repetition of 10 breaths with a one-minute interval between them. Total duration will be 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* with intermittent nonspecific CLBP for ≥12 weeks, with VAS between 3 to 7. All participants will be active at a recreational level, history of at least 12 weeks of NLBP, absence of radiculopathy or spinal damage due to tumors, stenosis, or fractures, and a minimum level of physical activity to be able to perform the exercises.

Exclusion Criteria:

* lumbar surgery experience,
* inflammatory spinal disease,
* spinal deformities,
* neurologic radiating pain

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Pain Level | Pre-intervention and 4 weeks Post-intervention
  Pain level will be assessed by the Numerical Rating Scale (NRS). The participants rated their pain on a defined 0-10 scale, where 0 is no pain, and 10 is the worst pain imaginable. NRS has different advantages, such as simplicity, reproducibility, and sensitivity to small changes in pain. NRS takes less than 1 min to complete and is a valid and reliable scale to measure pain intensity
Disability | Pre and 4 week post-intervention
  The disability due to NSLBP will be assessed using the Oswestry Disability Index (ODI), which is a self-administered questionnaire to evaluate the limitations of various daily living activities. The ODI is one of the most common scoring systems used for patients with LBP. The total score ranges from 0 to 100, where a higher score indicates a higher level of disability.
Flexibility | Pre and 4 weeks Post intervention
  The lumbar flexibility will be measured by Modified Schober test. The examiner puts his thumbs on the inferior margin of the subject's PSIS. An ink mark is drawn along the midline of the lumbar spine horizontal to the PSIS (lower landmark). While the examiner holds the tape firmly against the subject's skin, he marks a second line 15 cm above the original one (higher landmark). Then the subject is asked to do an active anterior flexion of the trunk without increasing the pain. The new distance between the lower and higher landmarks is then measured. The subject returns to the neutral position. The difference in the initial distance between the skin markings in the neutral position and the new measurements made in the flexion position is used to indicate the amount of lumbar flexion. Each therapist recorded measurements to the nearest mm

CONTACTS AND LOCATIONS:
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Background] Siglan U, Colak S. Effects of diaphragmatic and iliopsoas myofascial release in patients with chronic low back pain: A randomized controlled study. J Bodyw Mov Ther. 2023 Jan;33:120-127. doi: 10.1016/j.jbmt.2022.09.029. Epub 2022 Sep 29. PMID 36775506
- [Background] Otadi K, Nakhostin Ansari N, Sharify S, Fakhari Z, Sarafraz H, Aria A, Rasouli O. Effects of combining diaphragm training with electrical stimulation on pain, function, and balance in athletes with chronic low back pain: a randomized clinical trial. BMC Sports Sci Med Rehabil. 2021 Mar 4;13(1):20. doi: 10.1186/s13102-021-00250-y. PMID 33663607
- [Background] Masroor S, Tanwar T, Aldabbas M, Iram I, Veqar Z. Effect of Adding Diaphragmatic Breathing Exercises to Core Stabilization Exercises on Pain, Muscle Activity, Disability, and Sleep Quality in Patients With Chronic Low Back Pain: A Randomized Control Trial. J Chiropr Med. 2023 Dec;22(4):275-283. doi: 10.1016/j.jcm.2023.07.001. Epub 2023 Sep 2. PMID 38205226
- [Background] Oh YJ, Park SH, Lee MM. Comparison of Effects of Abdominal Draw-In Lumbar Stabilization Exercises with and without Respiratory Resistance on Women with Low Back Pain: A Randomized Controlled Trial. Med Sci Monit. 2020 Mar 17;26:e921295. doi: 10.12659/MSM.921295. PMID 32182226
- [Background] Gonzalez-Alvarez FJ, Valenza MC, Torres-Sanchez I, Cabrera-Martos I, Rodriguez-Torres J, Castellote-Caballero Y. Effects of diaphragm stretching on posterior chain muscle kinematics and rib cage and abdominal excursion: a randomized controlled trial. Braz J Phys Ther. 2016 Jun 16;20(5):405-411. doi: 10.1590/bjpt-rbf.2014.0169. PMID 27333481